CLINICAL TRIAL: NCT01926275
Title: Noninvasive Positive Pressure Ventilation Added Inspiratory Muscle Training in Severe Chronic Obstructive Pulmonary Disease
Brief Title: NPPV Added Inspiratory Muscle Training in Severe COPD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangzhou Institute of Respiratory Disease (Other)
Responsible Party: Principal Investigator, LuQian Zhou, Doctor, Guangzhou Institute of Respiratory Disease
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GZIRD-201308
Record Dates: First submitted 2013-08-14; First posted 2013-08-20 (Estimated); Last update posted 2013-08-20 (Estimated); Status verified 2013-08

CONDITIONS: Chronic Obstructive Pulmonary Disease; Hypercapnic Respiratory Failure
Keywords: COPD; Noninvasive Positive Pressure Ventilation; Respiratory Muscle Training
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Respiratory Insufficiency

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- NPPV+IMT (Experimental): noninvasive positive pressure ventilation and inspiratory muscle training
  Interventions: Device: NPPV; Device: IMT
- NPPV (Active Comparator): noninvasive positive pressure ventilation
  Interventions: Device: NPPV+IMT; Device: IMT
- IMT (Active Comparator): inspiratory muscle training
  Interventions: Device: NPPV+IMT; Device: NPPV
- LTOT (Placebo Comparator): Long time oxygen therapy
  Interventions: Device: NPPV+IMT; Device: NPPV; Device: IMT

INTERVENTIONS:
Device: NPPV+IMT — noninvasive positive pressure ventilation and inspiratory muscle training
  Arms: IMT; LTOT; NPPV
Device: NPPV — noninvasive positive pressure ventilation
  Arms: IMT; LTOT; NPPV+IMT
Device: IMT — inspiratory muscle training
  Arms: LTOT; NPPV; NPPV+IMT

SUMMARY:
The aim of this study is to determine whether noninvasive positive pressure ventilation with inspiratory muscle training can improve quality of life and respiratory muscle strength than noninvasive positive pressure ventilation or inspiratory muscle training alone.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 40-75 years, male or female.
2. Have spirometric evidence of COPD with an FEV1 of < 50% predicted and FEV1/FVC < 0.70, measured within the last 6 months (GOLD stage III and IV). Stable disease since 4 weeks or more prior to randomisation.
3. PCO2 of 7 kPa, combined with a pH of 7.35 or above. These gases must be measured after 30 minutes breathing room air in sitting position
4. No treatment with NPPV and respiratory muscle training in the last 8 weeks

Exclusion Criteria:

1. Smokers can be excluded;
2. Diseases of the lung or thorax besides COPD: OSA Advanced pulmonary fibrosis, advanced bronchiectases, active tuberculosis, post tuberculosis syndrome, pneumonia, severe kyphoscoliosis, tracheostoma, neuromuscular diseases, or any other disorder, which might result in elevated PCO2
3. Body mass index of 35 kg/m² or above. Severe cardiac disease, NYHA IV, instable angina, severe cardiac arrhythmia, especially of ventricular origin (atrial fibrillation is not an exclusion criterion).
4. Local derangement of the face, skin, tongue, upper airways, larynx and upper oesophagus.
5. Severe chronic diseases except COPD, hindering the patient to follow the schedule of this study

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2013-07; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Quality of life | Change from Baseline in quality of life at 8 weeks
  Severe Respiratory Insufficiency (SRI) Questionnaire and chronic obstructive pulmonary disease assessment test(CAT)

SECONDARY OUTCOMES:
respiratory muscle strength | Change from Baseline in respiratory muscle strength at 8 weeks
Dyspnea | Change from Baseline in dyspnea at 8 weeks
  baseline dyspnea index (BDI)and transition dyspnea index(TDI)
Walked distance in 6MWT | Change from Baseline in walked distance at 8 weeks
  Change from baseline in distance walked test 6-minute walk test at 8 week
Frequency of acute exacerbations of COPD | 8 week
Pulmonary function tests | Change from Baseline in pulmonary function tests at 8 weeks
Blood gases levels | Change from Baseline in blood gases levelsat 8 weeks
Sleep quality | Change from Baseline in sleep qualityat 8 weeks
  Epworth´s Sleepiness Scale
Length of hospital admission | 8 week
frequency of of hospital admission | 8 week

CONTACTS AND LOCATIONS:
Overall Officials: LuQian Zhou, Doctor, Principal Investigator — Guangzhou Institute of Respiratory Disease
Locations (1):
- Guangzhou Institute of Respiratory Disease, Guangzhou, Guangdong, China